CLINICAL TRIAL: NCT04770584
Title: Neural Correlates of Active Avoidance Learning and Their Interactions With Fear Extinction Mechanisms in PTSD Patients
Brief Title: Fear and Avoidance in PTSD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mohammed Milad, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-23-0495; R01MH123736 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional learning paradigm (Experimental): After the initial screening / baseline assessment visit, participants will undergo two Experimental Visits, which include participation in an emotional learning paradigm and an fMRI scan over the course of two consecutive days. Participants will be asked to look at pictures on a computer screen to measure physiological response physiological response (skin conductance response) and brain responses using a functional Magnetic Resonance Imaging (fMRI) machine. These two visits will be scheduled within a month from the baseline assessment visit.
  Interventions: Behavioral: Fear Conditioning; Other: Avoidance conditioning; Other: Pavlovian fear extinction learning; Other: Willingness to pay to avoid shock

INTERVENTIONS:
Behavioral: Fear Conditioning — Participants will be administered increasing intensities of mild electric shock via electrodes connected to the foot. New Biopac stimulators that can deliver higher shock intensity, provided participants agreement will be used to assure adequate conditioning levels. Stimulation is measures in milliamps (mA), and each delivered stimulation will be 0.5 seconds long (500 milliseconds). To colored (blue, red, & yellow) light stimuli (CS). The light stimulus is followed by a shock or no shock depending on color.
Other: Avoidance conditioning — Via button pressing. Only one stimulus-CS will enable control over experiencing the shock: the participant can press the button during the first 2 seconds of the light presentation to avoid the shock.
Other: Pavlovian fear extinction learning — After avoidance conditioning, the CS+ associated with avoidance responding appears with no button to press and no shock is administered.
Other: Willingness to pay to avoid shock — On the next day, participants receive a monetary stipend to use to pay to guarantee that they are not to receive any shocks if they press a button from the CS+. This and all previously described experimental phases noted above will occur inside of the fMRI scanner.

SUMMARY:
The purpose of this research study is to study how the brain learns to avoid certain stimuli or situations using an experimental paradigm. The big goal is to measure brain responses and subject's feelings and expectations when they are learning to actively avoid experimental stimuli, and how fear extinction learning and monetary cost can change how and when subjects are to avoid.

DETAILED DESCRIPTION:
This study aims to study the neural correlates of avoidance learning using a recently validated conditioning and active avoidance paradigm (CAAP). The overarching objective is to measure the neural correlates of active avoidance, and how fear extinction learning and monetary cost modulate these avoidance responses. Participants will include healthy controls (HC), trauma-exposed healthy controls (TEHC), and participants with post-traumatic stress disorder (PTSD). Avoidance is common and often hinders the progression and success of extinction-based exposure therapy in PTSD. The data to be gathered in this study will enable us to probe neural mechanisms of avoidance, extinction, and decision-making to avoid or not, in addition to understanding the impact of cost on avoidance decision-making. These data will provide a more integrated platform for the understanding of the mechanisms of avoidance in both trauma-exposed healthy controls and PTSD psychopathology, which has important implications for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 70 years of age
2. Female or Male
3. Inclusion Criteria: PTSD Subjects

   a. Diagnosis of current PTSD
4. Inclusion Criteria: Trauma-exposed healthy controls (TEHC)

   1. SCID diagnosis consistent with no current psychiatric disorders, and no current PTSD
   2. History of trauma exposure
5. Inclusion Criteria: Healthy controls (HC)

   1. SCID diagnosis consistent with no current psychiatric disorders ("Axis I" disorders).
   2. No history of trauma exposure
6. Willing and able to provide informed consent.

Exclusion Criteria for ALL subjects:

1. History of neurologic disease (e.g. tic disorder)
2. Current significant suicidal ideation, plan or intent or suicidal behavior in past 6 months based on CSSRS or Self-injurious behavior that involves suicidal intent, requires medical attention, or occurs daily
3. History of seizure or significant head trauma
4. History of the serious/significant psychiatric diagnosis ("Axis I" disorders)
5. Use of neuroleptics within one year prior to study
6. Current substance use (assessed by urine toxicology; positive urine toxicology screen for any substance, with the exception of THC). Per PI judgement and approval: if urine toxicology is positive for a substance, participant may be eligible to proceed with study provided their urine toxicology (or saliva test for THC) is negative at experimental visit(s)
7. Pregnancy (to be ruled out by urine ß-HCG)
8. Metallic implants or devices contraindicating magnetic resonance imaging
9. High risk of adverse emotional or behavioral reaction, and/or an inability to understand study procedures or the informed consent process

   Additional exclusion criteria for Trauma-exposed healthy controls (TEHC) group and Healthy controls (HC) group:
10. Current psychiatric diagnosis ("Axis I" diagnoses)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Skin Conductance Response (SCR) | Experimental Day 1, Experimental Day 2
  Skin Conductance Response (SCR) assesses the stress/seat level, or level of anxiety in a particular moment, or in response to a specific cue. SCR will be reported in microsiemens.
Functional MRI (fMRI) responses | Experimental Day 1, Experimental Day 2
  fMRI data, including blood-oxygen-level-dependent (BOLD) responses, is used in neuroimaging studies assess neural correlate activations and observe the increase/decrease in activation of a particular brain area in response to a specific cue.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milad, PhD, Principal Investigator — The University of Texas Health Science Center at Houston (UTHealth Houston)
Locations (1):
- UTHealth Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access and give upon reasonable request. Requests should be directed to Mohammed.R.Milad@uth.tmc.edu. To gain access, data requestors will need to sign a data access agreement.